CLINICAL TRIAL: NCT03960489
Title: A Phase 1 Crossover Study to Assess the Relative Bioavailability of Roxadustat Following a Single Dose of Pediatric Azo Dye-free Tablet and Pediatric Azo Dye-free Mini-tablet (Solid and Suspension) Compared to a Single Dose of Azo Dye-containing Tablet in Healthy Adult Subjects
Brief Title: A Study to Assess the Relative Bioavailability of Roxadustat Following a Single Dose of Pediatric Azo Dye-free Tablet Formulation and Pediatric Azo Dye-free Mini-tablet Formulation Compared to a Single Dose of Azo Dye-containing Tablet Formulation in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1517-CL-1001; 2018-002924-18 (EudraCT Number)
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Healthy Adult Subjects
Keywords: Pharmacokinetics; Tolerability; Safety; ASP1517; Roxadustat
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment Sequence 1 (ABCD) (Experimental): Participants will receive single dose of 100 mg roxadustat pediatric azo dye-free tablet (A), orally on day 1 in period 1 followed by 100 mg roxadustat pediatric azo dye-free mini-tablet suspension (B), orally on day 1 in period 2 followed by 100 mg roxadustat pediatric azo dye-free mini-tablet solid (C), orally on day 1 in period 3 followed by 100 mg roxadustat azo dye-containing tablet (D), orally on day 1 in period 4. Each period will be of 6 days. A washout period of 7 days will be included between each period.
  Interventions: Drug: Roxadustat
- Treatment Sequence 2 (BDAC) (Experimental): Participants will receive 100 mg roxadustat pediatric azo dye-free mini-tablet suspension (B), orally on day 1 in period 1 followed by single dose of 100 mg roxadustat azo dye-containing tablet (D), orally on day 1 in period 2 followed by 100 mg roxadustat pediatric azo dye-free tablet (A), orally on day 1 in period 3 followed by 100 mg roxadustat pediatric azo dye-free mini-tablet solid (C), orally on day 1 in period 4. Each period will be of 6 days. A washout period of 7 days will be included between each period.
  Interventions: Drug: Roxadustat
- Treatment Sequence 3 (CADB) (Experimental): Participants will receive single dose of 100 mg roxadustat pediatric azo dye-free mini-tablet solid (C), orally on day 1 in period 1 followed by 100 mg roxadustat pediatric azo dye-free tablet (A), orally on day 1 in period 2 followed by 100 mg roxadustat azo dye-containing tablet (D), orally on day 1 in period 3 followed by 100 mg roxadustat pediatric azo dye-free mini-tablet suspension (B), orally on day 1 in period 4. Each period will be of 6 days. A washout period of 7 days will be included between each period.
  Interventions: Drug: Roxadustat
- Treatment Sequence 4 (DCBA) (Experimental): Participants will receive single dose of 100 mg roxadustat azo dye-containing tablet (D), orally on day 1 in period 1 followed by 100 mg roxadustat pediatric azo dye-free mini-tablet solid (C), orally on day 1 in period 2 followed by 100 mg roxadustat pediatric azo dye-free mini-tablet suspension (B), orally on day 1 in period 3 followed by 100 mg of roxadustat pediatric azo dye-free tablet (A), orally on day 1 in period 4. Each period will be of 6 days. A washout period of 7 days will be included between each period.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Participants will receive single dose of 100 mg azo dye free tablet or mini tablet suspension or solid mini tablet or dye containing tablet.
  Other Names: ASP1517

SUMMARY:
The purpose of the study is to assess the relative bioavailability of single doses of 100 mg roxadustat pediatric azo dye-free tablet and 100 mg roxadustat pediatric azo dye-free mini-tablet solid and suspension (new formulations) compared to 100 mg roxadustat azo dye-containing tablet (reference formulation) under fasting conditions in healthy male and female adult participants.

This study will also evaluate the safety and tolerability of single doses of 100 mg roxadustat pediatric azo dye-free tablet and 100 mg roxadustat pediatric azo dye-free mini-tablet solid and suspension (new formulations) and a single dose of 100 mg roxadustat azo dye-containing tablet (reference formulation) under fasting conditions in healthy male and female adult participants.

DETAILED DESCRIPTION:
This is a 4-period, 4-sequence single dose crossover study. Each participant will participate in 4 treatment periods separated by a washout of at least 7 days between study drug administrations in each period. Participants will be randomized to 1 of 4 sequences.

Participants will be screened for up to 21 days prior to study drug administration on day 1 of period 1. Eligible participants will be admitted to the clinical unit on day -1 of each period and will be residential for 5 days/4 nights.

Participants will receive a single dose of 100 mg roxadustat pediatric azo dye-free tablet, 100 mg roxadustat pediatric azo dye-free mini-tablet (suspension), 100 mg roxadustat pediatric azo dye-free mini-tablet (solid) (new formulations) or 100 mg roxadustat azo dye-containing tablet (reference formulation) under fasting conditions on day 1 of each period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 18.5 to 30.0 kg/m2, inclusive and weighs at least 50 kg at screening.
* A female subject is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP), or
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 28 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period and for 28 days after the final study drug administration.
* A male subject with female partner(s) of childbearing potential must agree to use contraception during the treatment period and for at least 28 days after the final study drug administration.
* A male subject must not donate sperm during the treatment period and for at least 28 days after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner(s) is (are) breastfeeding throughout the study period and for 28 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has received any investigational study drug within 28 days or 5 half lives, whichever is longer, prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to roxadustat or any components of the formulation used.
* Subject has had previous exposure with roxadustat.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, gamma-glutamyl transferase and total bilirubin [TBL]) above the upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to study drug administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality of the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or on day -1.
* Subject has a mean pulse < 50 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional measurement in triplicate can be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) of > 430 msec (for male subjects) and > 450 msec (for female subjects) on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, calcium and iron supplements, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day), topical dermatological products, including corticosteroid products, hormonal contraceptives and hormone replacement therapy.
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine-containing products in the past 6 months prior to screening.
* Subject has a history of drinking more than 24 g/day of alcohol (10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) (> 12 g/day of alcohol for female subjects) within 3 months prior to day -1 or the subject tests positive for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -1.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) within 3 months prior to day -1.
* Subject has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Subject has consumed grapefruit, Seville oranges, grapefruit-containing products or Seville orange-containing products within 72 hours prior to day -1.
* Subject has had significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day -1.
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis B core antibodies, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Subject is an employee of Astellas or the clinical site.
* Subject is a vulnerable subject (e.g., subject kept in detention, protected adult under guardianship/trusteeship, soldier or committed to an institution by governmental or juridical order).
* Subject has abnormal renal function, indicated by creatinine above the ULN or chronic kidney disease epidemiology collaboration based estimated glomerular filtration rate (eGFR) < 90 mL/min on day 1. In such a case, the assessment may be repeated once.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time of Dosing Extrapolated to Time Infinity (AUCinf) for Roxadustat | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  AUCinf is defined as area under the plasma concentration versus time curve from time of dosing (pre-dose) to extrapolated infinite time (0-inf).
Area Under the Concentration-Time Curve From the Time of Dosing to Last Measurable Concentration (AUClast) for Roxadustat | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  AUClast is defined as area under the plasma concentration time-curve from time of dosing to the last measured concentration.
Pharmacokinetics (PK) of Maximum Observed Concentration of Roxadustat | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  Maximum observed concentration (Cmax) will be reported.

SECONDARY OUTCOMES:
Percentage of the Area Under the Concentration-Time Curve From the Time of Dosing to Time infinity due to Extrapolation From the Last Measurable Concentration to Time Infinity (AUCinf[%extrap]) for Roxadustat | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  AUC%extrap is defined as the percentage of AUC [0-∞] obtained by forward extrapolation. It will be calculated as (AUC [0-∞] minus AUClast)*100/ AUC [0-∞], where AUC [0-∞] = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-∞) and AUClast is area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration.
Apparent Total Systemic Clearance of Roxadustat After Extravascular Dosing (CL/F) | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Terminal Elimination Half-life (t1/2) of Roxadustat | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time to Reach Maximum Concentration (tmax) of Roxadustat | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  Time to reach maximum concentration of roxadustat following drug administration will be reported.
Time Prior to the Time Corresponding to the First Measurable (nonzero) Concentration (tlag) of Roxadustat | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  Tlag is defined as the time prior to the time corresponding to the first measurable concentration.
Apparent Volume of Distribution During the Terminal Elimination Phase After Extravascular Dosing (Vz/F) of Roxadustat | Predose (0 hour), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose on day 1
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Number of Participants With Treatment-Emergent Adverse Event (TEAEs) | From first dose of study drug up to end of study visit (up to 54 days)
  An AE is defined as any untoward medical occurrence in a participant who will be given the study drug or who has undergone study procedures and did not necessarily has a causal relationship with this treatment. An AE could therefore be any unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A treatment-emergent adverse event is defined as an adverse event with onset at any time from dosing until the last scheduled procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Site DE49001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.